CLINICAL TRIAL: NCT05766384
Title: Hyperpolarized 129Xe MRI to Identify Structural Determinants of Low Lung Function and Respiratory Symptoms in Young Adults From the Lung Health Cohort
Brief Title: Hyperpolarized 129Xe MRI Lung Health Cohort
Acronym: XeLHC
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Johns Hopkins University (Other); University of Iowa (Other); Duke University (Other); University of Illinois at Chicago (Other); Baylor College of Medicine (Other); Temple University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Peter J. Niedbalski, PhD, Research Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY00160099
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Xenon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Inhaled hyperpolarized 129Xe used as a signal agent for MRI of the lungs.
  Other Names: Xenon, 129Xe, HP Xenon

SUMMARY:
A subset of young adults participating in the American Lung Association (ALA) Lung Health Cohort (LHC) will be imaged using Hyperpolarized 129Xe MRI to assess lung structure and function. Images will be used to improve the understanding of lung health and early lung abnormalities that may lead to chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Is enrolled in the American Lung Association Lung Health Cohort Study.
* Has completed CT imaging for the LHC study within 2 years of the scheduled Xe-MRI date.

Exclusion Criteria:

* Pacemaker, internal defibrillator or other implanted electronic devices or any standard MRI contraindications (e.g., claustrophobia, > 140 cm shoulder circumference, dependent on weight distribution).
* Is pregnant or breastfeeding
* Oxygen saturation (SpO2) <88% on room air or with supplemental oxygen.

Ages: 25 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Participants enrolled in the Lung Health Cohort at participating Airways Clinical Research Centers. The investigators target to enroll approximately 50% females and enroll approximately 1/3 low socioeconomic status (SES) participants, 1/3 middle SES, and 1/3 high SES. The target for the population demographics is to match those of the larger, LHC parent study.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Xe-MRI Apparent Diffusion Coefficient | At baseline imaging timepoint
  Correlation of Xe-MRI with FEV1/FVC and other measures of lung function

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Illinois-Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Duke University, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified imaging data will be made available to researchers by publishing on a data sharing site. Images will be made available upon completion of the study and publication of the summary paper.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available indefinitely upon completion of the study (anticipated 3/31/2028)